CLINICAL TRIAL: NCT00730535
Title: Exploring Predictors of Symptoms Relapse After Discontinuation of Successful Treatment With a Tolterodine Prolonged Release Capsules (4 mg, Once Daily) in Overactive Bladder Patients: A Prospective Randomized Multicenter Trial
Brief Title: Exploring Predictors of Symptoms Relapse After Discontinuation of Treatment in Overactive Bladder (OAB) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KYU-SUNG LEE (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor-Investigator, KYU-SUNG LEE, professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-08-069
Record Dates: First submitted 2008-08-07; First posted 2008-08-08 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2011-04

CONDITIONS: Overactive Bladder
Keywords: Overactive bladder, Tolterodine,Symptoms Relapse, Predictor
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tolterodine 1 (Experimental)
  Interventions: Drug: Tolterodine
- Toterodine 3 (Experimental)
  Interventions: Drug: Tolterodine
- Tolterodine 6 (Experimental)
  Interventions: Drug: Tolterodine 6

INTERVENTIONS:
Drug: Tolterodine — Extended release tolterodine tartrate 4 mg, once daily, for 1 months
  Other Names: Detrusitol ER 4mg
  Arms: Tolterodine 1
Drug: Tolterodine — Extended release tolterodine tartrate 4 mg, once daily, for 3 months
  Other Names: Detrusitol ER 4mg
  Arms: Toterodine 3
Drug: Tolterodine 6 — Extended release tolterodine tartrate 4 mg, once daily, for 6 months
  Other Names: Detrusitol ER 4mg
  Arms: Tolterodine 6

SUMMARY:
This is a Phase IV, prospective, randomized, multi-center study to find risk factors of OAB symptoms relapse in patients who showed therapeutic benefits after 1, 3, or 6 months of treatment with Tolterodine SR and who then discontinued these antimuscarinics for 3 month.

Patients who have OAB symptoms for 6 or more than 6 months and who show successful treatment response to 1 month of treatment with Tolterodine SR 4mg will be enrolled and randomized to 1, 3 or 6 months of treatment group. After completion of the treatment, subjects will be evaluated for changes in OAB symptoms and retreatment rate will be assessed.

DETAILED DESCRIPTION:
Primary Objective:

* To investigate the risk factors of OAB symptom relapse and retreatment in patients who showed therapeutic benefits after 1, 3 or 6 months of treatment with Tolterodine SR and who then discontinued these antimuscarinics for 3 month.

Secondary Objective:

* To investigate the change of the patient perception and quality of life after antimuscarinic discontinuation
* To find the rate of patients who have OAB symptom relapse.
* To find the risk factors of patients who want retreatment.
* To find the rate of patients who want retreatment.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18≤and ≤80 years
2. Symptoms of urinary urgency (defined as a level of 3 to 5 in a 5 point Urinary Sensation Scale) over 2 times per day
3. Symptoms of urinary frequency (≥ 8 micturitions per 24 hours) as verified by baseline micturition diary.
4. Symptoms of overactive bladder, including urinary urge incontinence, urgency and/or frequency for ≥6 months.
5. Ability and willingness to correctly complete the micturition diary and questionnaire
6. Capable of understanding and having signed the informed consent form after full discussion of the research nature of the treatment and its risks and benefits

Exclusion Criteria:

1. Clinical significant stress incontinence as determined by the investigator and confirmed for female patients by a cough provocation test
2. An average volume voided of > 200 ml per micturition as verified on the baseline micturition diary
3. Total daily urine volume of > 3000 ml as verified on the baseline micturition diary
4. Significant hepatic or renal disease, defined as having twice the upper limit of the reference ranges for serum concentrations of aspartate aminotransferase (AST [SGOT]), alanine aminotransferase (ALT [SGPT]), alkaline phosphatase or creatinine
5. Any condition that is a contraindication for anticholinergic treatment, including uncontrolled narrow-angled glaucoma, urinary retention or gastric retention
6. Symptomatic acute urinary tract infection (UTI) during the run-in period
7. Recurrent UTIs defined as having been treated for symptomatic UTIs > 4 times in the last year
8. Diagnosed or suspected interstitial cystitis
9. Uninvestigated hematuria or hematuria secondary to malignant disease.
10. Clinically significant bladder outlet obstruction defined by clinical symptoms and investigator's opinion according to local standard of care
11. Patients with marked cystocele or other clinically significant pelvic prolapse.
12. On an unstable dosage of any drug with anticholinergic side effects, or expected to start such treatment during the study
13. Receipt of any electrostimulation or bladder training within the 14 days before the start of tolterodine SR, or expected to start such treatment during the study
14. Use of any other drugs for the treatment of overactive bladder (e.g. anticholinergics except tolterodine) within the 14 days before the start of tolterodine SR, or expected to start such treatment during the study
15. An indwelling catheter or practicing intermittent self-catheterization
16. Use of any investigational drug within 2 months preceding the start of the study
17. Patients with chronic constipation or history of severe constipation
18. Pregnant or nursing women
19. Sexually active females of childbearing potential not using reliable contraception for at least 1 month prior to study start and not agreeing to use such methods during the entire study period and for at least 1 month thereafter. Reliable contraceptive methods are defined as intrauterine devices (IUDs), combination type contraceptive pills, hormonal implants, double barrier method, injectable contraceptives and surgical procedures (tubal ligation or vasectomy).
20. Patients who have bladder cancer
21. Treatment with potent CYP3A4 inhibitors, such as cyclosporine, vinblastine, macrolide antibiotics (e.g. erythromycin, clarithromycin, azithromycin) or antifungal agents (e.g. ketoconazole, itraconazole, micronazole).
22. Any other condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2006-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Risk factors and relapse rate of the OAB symptoms after drug discontinuation | from baseline (treatment completion) to 1, 3 month after drug discontinuation

SECONDARY OUTCOMES:
Micturition diary efficacy parameters | from baseline (treatment completion) to 1, 3 month after drug discontinuation
Quality of life parameters: change in total score and subscale scores of OAB-questionnaire | from baseline (treatment completion) to 1, 3 month after drug discontinuation
Patient perceptions: change in patient perception of urgency, change in patient perception of bladder condition and percentage of patients who wants retreatment | from baseline (treatment completion) to 1, 3 month after drug discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (4):
- South Korea (4):
  - Samsung Medical Center, Irwon-dong, Seoul
  - Holy Family Hospital, The Catholic University of Korea, Gyeonggi-do
  - Asan Medical Center, Ulsan College of Medicine, Seoul
  - Seoul National University Hospital, Seoul